CLINICAL TRIAL: NCT04894409
Title: Evaluation of Silver Nanoparticles as an Oropharyngeal Product (Mouthwash) and Nasal Hygiene, by Health Personnel Working at the Tijuana General Hospital Exposed to Patients Diagnosed With Atypical Pneumonia Caused by SARS-CoV-2
Brief Title: Evaluation of Silver Nanoparticles for the Prevention of COVID-19
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cluster de Bioeconomia de Baja California, A.C (Other)
Collaborators: Bionag SAPI de CV (Unknown); General Hospital Tijuana (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CONBIOETICA-02-CEI-001-20170
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: Silver nanoparticles; SARS-CoV-2; COVID-19; Infection control
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Eligible participants for the in vivo study were randomized using a computer generated block scheme and stratified according to duty position, work shifts and the area/department of the service at General Tijuana Hospital. Individuals from experimental group were provided with a 50 mL spray bottle containing AgNPs solution with 1 wt% concentration (0.6 mg/mL metallic silver). Participants were instructed to mix 4 to 6 spray shots (corresponding to volume ~ 0.5 mL) of this solution with 20 mL of water and to gargle with obtained solution for 15 to 30 seconds at least 3 times a day, also nasal lavages on the inner part of the nasal alae and nasal passage with the same solution using a cotton swap twice a day. As a second option, participants were instructed to cover evenly the oral cavity with the direct 1 to 2 spray shots of solution without its previous dilution in water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental group was instructed to do mouthwash and nose rinse with the AgNPs solution.
  Interventions: Device: Mouthwash and nose rinse with the AgNPs solution
- Control group (Active Comparator): The "control" group was instructed to do mouthwashes and nose rinse in a conventional way.
  Interventions: Device: Mouthwashes and nose rinse in a conventional way

INTERVENTIONS:
Device: Mouthwash and nose rinse with the AgNPs solution — The "experimental" group was instructed to do mouthwash and nose rinse with the AgNPs solution for the prevention of SARS-CoV-2 infection in health workers
  Arms: Experimental group
Device: Mouthwashes and nose rinse in a conventional way — The control group was instructed to do mouthwashes and nose rinse in a conventional way
  Arms: Control group

SUMMARY:
In this research, silver nanoparticles (AgNPs) were tested in vitro and shown to have an inhibitory effect on SARS-CoV-2 infection in cultured cells. Subsequently, the investigators assessed the effects of mouthwash and nose rinse with ARGOVIT® silver nanoparticles (AgNPs), in the prevention of SARS-CoV-2 contagion in health workers consider as high-risk group of acquiring the infection in the General Tijuana Hospital, Mexico, a hospital for the exclusive recruitment of patients diagnosed with COVID-19.

DETAILED DESCRIPTION:
SARS-CoV-2 infection in hospital areas is of a particular concern, since the close interaction between health care personnel and patients diagnosed with COVID-19, which allows virus to be easily spread between them and subsequently to their families and communities. Preventing SARS-CoV-2 infection among healthcare personnel is essential to reduce the frequency of infections and outbreaks during the pandemic. In a first step, silver nanoparticles (AgNPs) were tested in vitro to determine an inhibitory effect on SARS-CoV-2 infection in cultured cells. Subsequently, the investigators assess the effects of mouthwash and nose rinse with ARGOVIT® silver nanoparticles (AgNPs), in the prevention of SARS-CoV-2 contagion in health workers consider as high-risk group of acquiring the infection in the General Tijuana Hospital, Mexico, a hospital for the exclusive recruitment of patients diagnosed with COVID-19. The investigators present a prospective randomized study of 231 participants that was carried out for 9 weeks (during the declaration of a pandemic). The "experimental" group was instructed to do mouthwash and nose rinse with the AgNPs solution; the "control" group was instructed to do mouthwashes and nose rinse in a conventional way.

ELIGIBILITY:
Inclusion Criteria:

* Men and women health workers in the General Tijuana Hospital, Mexico who works in high-risk areas with direct contact with patients infected and diagnosed with COVID-19.

Exclusion Criteria:

* persons with history of hypersensitivity to silver (rashes and other contraindications),
* a history of SARS-CoV-2 infection in the three months prior to the start of the study, any respiratory distress,
* and refusal to sign the informed consent.

Ages: 20 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Incidence of SARS-CoV-2 infection in the experimental group. | 9 weeks
  Percentage of participants infected of SARS-CoV-2 in the experimental group.
Incidence of SARS-CoV-2 infection in the control group. | 9 weeks
  Percentage of participants infected of SARS-CoV-2 in the control group.

SECONDARY OUTCOMES:
Number of participants with adverse reactions by AgNPs. | 9 weeks
  Number of participants with adverse reactions by performing mouthwash and nose rinse with AgNPs.

CONTACTS AND LOCATIONS:
Locations (1):
- Tijuana General Hospital, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lan FY, Wei CF, Hsu YT, Christiani DC, Kales SN. Work-related COVID-19 transmission in six Asian countries/areas: A follow-up study. PLoS One. 2020 May 19;15(5):e0233588. doi: 10.1371/journal.pone.0233588. eCollection 2020. PMID 32428031
- [Background] Wong SCY, Kwong RT, Wu TC, Chan JWM, Chu MY, Lee SY, Wong HY, Lung DC. Risk of nosocomial transmission of coronavirus disease 2019: an experience in a general ward setting in Hong Kong. J Hosp Infect. 2020 Jun;105(2):119-127. doi: 10.1016/j.jhin.2020.03.036. Epub 2020 Apr 4. PMID 32259546
- [Background] Wee LE, Hsieh JYC, Phua GC, Tan Y, Conceicao EP, Wijaya L, Tan TT, Tan BH. Respiratory surveillance wards as a strategy to reduce nosocomial transmission of COVID-19 through early detection: The experience of a tertiary-care hospital in Singapore. Infect Control Hosp Epidemiol. 2020 Jul;41(7):820-825. doi: 10.1017/ice.2020.207. Epub 2020 May 8. PMID 32381147
- [Background] Ho HJ, Zhang ZX, Huang Z, Aung AH, Lim WY, Chow A. Use of a Real-Time Locating System for Contact Tracing of Health Care Workers During the COVID-19 Pandemic at an Infectious Disease Center in Singapore: Validation Study. J Med Internet Res. 2020 May 26;22(5):e19437. doi: 10.2196/19437. PMID 32412416
- [Background] Jeon S, Ko M, Lee J, Choi I, Byun SY, Park S, Shum D, Kim S. Identification of Antiviral Drug Candidates against SARS-CoV-2 from FDA-Approved Drugs. Antimicrob Agents Chemother. 2020 Jun 23;64(7):e00819-20. doi: 10.1128/AAC.00819-20. Print 2020 Jun 23. PMID 32366720
- [Background] Park SJ, Yu KM, Kim YI, Kim SM, Kim EH, Kim SG, Kim EJ, Casel MAB, Rollon R, Jang SG, Lee MH, Chang JH, Song MS, Jeong HW, Choi Y, Chen W, Shin WJ, Jung JU, Choi YK. Antiviral Efficacies of FDA-Approved Drugs against SARS-CoV-2 Infection in Ferrets. mBio. 2020 May 22;11(3):e01114-20. doi: 10.1128/mBio.01114-20. PMID 32444382
- [Background] Logunov DY, Dolzhikova IV, Shcheblyakov DV, Tukhvatulin AI, Zubkova OV, Dzharullaeva AS, Kovyrshina AV, Lubenets NL, Grousova DM, Erokhova AS, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Egorova DA, Shmarov MM, Nikitenko NA, Gushchin VA, Smolyarchuk EA, Zyryanov SK, Borisevich SV, Naroditsky BS, Gintsburg AL; Gam-COVID-Vac Vaccine Trial Group. Safety and efficacy of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine: an interim analysis of a randomised controlled phase 3 trial in Russia. Lancet. 2021 Feb 20;397(10275):671-681. doi: 10.1016/S0140-6736(21)00234-8. Epub 2021 Feb 2. PMID 33545094
- [Background] Zhu FC, Guan XH, Li YH, Huang JY, Jiang T, Hou LH, Li JX, Yang BF, Wang L, Wang WJ, Wu SP, Wang Z, Wu XH, Xu JJ, Zhang Z, Jia SY, Wang BS, Hu Y, Liu JJ, Zhang J, Qian XA, Li Q, Pan HX, Jiang HD, Deng P, Gou JB, Wang XW, Wang XH, Chen W. Immunogenicity and safety of a recombinant adenovirus type-5-vectored COVID-19 vaccine in healthy adults aged 18 years or older: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2020 Aug 15;396(10249):479-488. doi: 10.1016/S0140-6736(20)31605-6. Epub 2020 Jul 20. PMID 32702299
- [Background] Folegatti PM, Ewer KJ, Aley PK, Angus B, Becker S, Belij-Rammerstorfer S, Bellamy D, Bibi S, Bittaye M, Clutterbuck EA, Dold C, Faust SN, Finn A, Flaxman AL, Hallis B, Heath P, Jenkin D, Lazarus R, Makinson R, Minassian AM, Pollock KM, Ramasamy M, Robinson H, Snape M, Tarrant R, Voysey M, Green C, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of the ChAdOx1 nCoV-19 vaccine against SARS-CoV-2: a preliminary report of a phase 1/2, single-blind, randomised controlled trial. Lancet. 2020 Aug 15;396(10249):467-478. doi: 10.1016/S0140-6736(20)31604-4. Epub 2020 Jul 20. PMID 32702298
- [Background] Jackson LA, Anderson EJ, Rouphael NG, Roberts PC, Makhene M, Coler RN, McCullough MP, Chappell JD, Denison MR, Stevens LJ, Pruijssers AJ, McDermott A, Flach B, Doria-Rose NA, Corbett KS, Morabito KM, O'Dell S, Schmidt SD, Swanson PA 2nd, Padilla M, Mascola JR, Neuzil KM, Bennett H, Sun W, Peters E, Makowski M, Albert J, Cross K, Buchanan W, Pikaart-Tautges R, Ledgerwood JE, Graham BS, Beigel JH; mRNA-1273 Study Group. An mRNA Vaccine against SARS-CoV-2 - Preliminary Report. N Engl J Med. 2020 Nov 12;383(20):1920-1931. doi: 10.1056/NEJMoa2022483. Epub 2020 Jul 14. PMID 32663912
- [Background] Keech C, Albert G, Cho I, Robertson A, Reed P, Neal S, Plested JS, Zhu M, Cloney-Clark S, Zhou H, Smith G, Patel N, Frieman MB, Haupt RE, Logue J, McGrath M, Weston S, Piedra PA, Desai C, Callahan K, Lewis M, Price-Abbott P, Formica N, Shinde V, Fries L, Lickliter JD, Griffin P, Wilkinson B, Glenn GM. Phase 1-2 Trial of a SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine. N Engl J Med. 2020 Dec 10;383(24):2320-2332. doi: 10.1056/NEJMoa2026920. Epub 2020 Sep 2. PMID 32877576
- [Background] Guan Y, Zheng BJ, He YQ, Liu XL, Zhuang ZX, Cheung CL, Luo SW, Li PH, Zhang LJ, Guan YJ, Butt KM, Wong KL, Chan KW, Lim W, Shortridge KF, Yuen KY, Peiris JS, Poon LL. Isolation and characterization of viruses related to the SARS coronavirus from animals in southern China. Science. 2003 Oct 10;302(5643):276-8. doi: 10.1126/science.1087139. Epub 2003 Sep 4. PMID 12958366
- [Background] Zaki AM, van Boheemen S, Bestebroer TM, Osterhaus AD, Fouchier RA. Isolation of a novel coronavirus from a man with pneumonia in Saudi Arabia. N Engl J Med. 2012 Nov 8;367(19):1814-20. doi: 10.1056/NEJMoa1211721. Epub 2012 Oct 17. PMID 23075143
- [Background] Ren LL, Wang YM, Wu ZQ, Xiang ZC, Guo L, Xu T, Jiang YZ, Xiong Y, Li YJ, Li XW, Li H, Fan GH, Gu XY, Xiao Y, Gao H, Xu JY, Yang F, Wang XM, Wu C, Chen L, Liu YW, Liu B, Yang J, Wang XR, Dong J, Li L, Huang CL, Zhao JP, Hu Y, Cheng ZS, Liu LL, Qian ZH, Qin C, Jin Q, Cao B, Wang JW. Identification of a novel coronavirus causing severe pneumonia in human: a descriptive study. Chin Med J (Engl). 2020 May 5;133(9):1015-1024. doi: 10.1097/CM9.0000000000000722. PMID 32004165
- [Background] Jaume M, Yip MS, Cheung CY, Leung HL, Li PH, Kien F, Dutry I, Callendret B, Escriou N, Altmeyer R, Nal B, Daeron M, Bruzzone R, Peiris JS. Anti-severe acute respiratory syndrome coronavirus spike antibodies trigger infection of human immune cells via a pH- and cysteine protease-independent FcgammaR pathway. J Virol. 2011 Oct;85(20):10582-97. doi: 10.1128/JVI.00671-11. Epub 2011 Jul 20. PMID 21775467
- [Background] Li L, Wo J, Shao J, Zhu H, Wu N, Li M, Yao H, Hu M, Dennin RH. SARS-coronavirus replicates in mononuclear cells of peripheral blood (PBMCs) from SARS patients. J Clin Virol. 2003 Dec;28(3):239-44. doi: 10.1016/s1386-6532(03)00195-1. PMID 14522061
- [Background] Gu J, Gong E, Zhang B, Zheng J, Gao Z, Zhong Y, Zou W, Zhan J, Wang S, Xie Z, Zhuang H, Wu B, Zhong H, Shao H, Fang W, Gao D, Pei F, Li X, He Z, Xu D, Shi X, Anderson VM, Leong AS. Multiple organ infection and the pathogenesis of SARS. J Exp Med. 2005 Aug 1;202(3):415-24. doi: 10.1084/jem.20050828. Epub 2005 Jul 25. PMID 16043521
- [Background] Ochoa-Meza AR, Alvarez-Sanchez AR, Romo-Quinonez CR, Barraza A, Magallon-Barajas FJ, Chavez-Sanchez A, Garcia-Ramos JC, Toledano-Magana Y, Bogdanchikova N, Pestryakov A, Mejia-Ruiz CH. Silver nanoparticles enhance survival of white spot syndrome virus infected Penaeus vannamei shrimps by activation of its immunological system. Fish Shellfish Immunol. 2019 Jan;84:1083-1089. doi: 10.1016/j.fsi.2018.10.007. Epub 2018 Oct 30. PMID 30389645
- [Background] Borrego B, Lorenzo G, Mota-Morales JD, Almanza-Reyes H, Mateos F, Lopez-Gil E, de la Losa N, Burmistrov VA, Pestryakov AN, Brun A, Bogdanchikova N. Potential application of silver nanoparticles to control the infectivity of Rift Valley fever virus in vitro and in vivo. Nanomedicine. 2016 Jul;12(5):1185-92. doi: 10.1016/j.nano.2016.01.021. Epub 2016 Mar 10. PMID 26970026
- [Background] Salleh A, Naomi R, Utami ND, Mohammad AW, Mahmoudi E, Mustafa N, Fauzi MB. The Potential of Silver Nanoparticles for Antiviral and Antibacterial Applications: A Mechanism of Action. Nanomaterials (Basel). 2020 Aug 9;10(8):1566. doi: 10.3390/nano10081566. PMID 32784939
- [Background] Cardoso VS, Quelemes PV, Amorin A, Primo FL, Gobo GG, Tedesco AC, Mafud AC, Mascarenhas YP, Correa JR, Kuckelhaus SA, Eiras C, Leite JR, Silva D, dos Santos Junior JR. Collagen-based silver nanoparticles for biological applications: synthesis and characterization. J Nanobiotechnology. 2014 Sep 17;12:36. doi: 10.1186/s12951-014-0036-6. PMID 25223611
- [Background] Jeremiah SS, Miyakawa K, Morita T, Yamaoka Y, Ryo A. Potent antiviral effect of silver nanoparticles on SARS-CoV-2. Biochem Biophys Res Commun. 2020 Nov 26;533(1):195-200. doi: 10.1016/j.bbrc.2020.09.018. Epub 2020 Sep 11. PMID 32958250
- [Background] Schwartz J, King CC, Yen MY. Protecting Healthcare Workers During the Coronavirus Disease 2019 (COVID-19) Outbreak: Lessons From Taiwan's Severe Acute Respiratory Syndrome Response. Clin Infect Dis. 2020 Jul 28;71(15):858-860. doi: 10.1093/cid/ciaa255. PMID 32166318
- [Background] Casale M, Rinaldi V, Sabatino L, Moffa A, Ciccozzi M. Could nasal irrigation and oral rinse reduce the risk for COVID-19 infection? Int J Immunopathol Pharmacol. 2020 Jan-Dec;34:2058738420941757. doi: 10.1177/2058738420941757. PMID 32799596
- [Background] Singh S, Sharma N, Singh U, Singh T, Mangal DK, Singh V. Nasopharyngeal wash in preventing and treating upper respiratory tract infections: Could it prevent COVID-19? Lung India. 2020 May-Jun;37(3):246-251. doi: 10.4103/lungindia.lungindia_241_20. PMID 32367847
- [Background] To KK, Tsang OT, Yip CC, Chan KH, Wu TC, Chan JM, Leung WS, Chik TS, Choi CY, Kandamby DH, Lung DC, Tam AR, Poon RW, Fung AY, Hung IF, Cheng VC, Chan JF, Yuen KY. Consistent Detection of 2019 Novel Coronavirus in Saliva. Clin Infect Dis. 2020 Jul 28;71(15):841-843. doi: 10.1093/cid/ciaa149. PMID 32047895
- [Background] Khan MM, Parab SR, Paranjape M. Repurposing 0.5% povidone iodine solution in otorhinolaryngology practice in Covid 19 pandemic. Am J Otolaryngol. 2020 Sep-Oct;41(5):102618. doi: 10.1016/j.amjoto.2020.102618. Epub 2020 Jun 18. PMID 32574894
- [Background] Butowt R, Bilinska K. SARS-CoV-2: Olfaction, Brain Infection, and the Urgent Need for Clinical Samples Allowing Earlier Virus Detection. ACS Chem Neurosci. 2020 May 6;11(9):1200-1203. doi: 10.1021/acschemneuro.0c00172. Epub 2020 Apr 13. PMID 32283006
- [Background] Uskokovic V. Why have nanotechnologies been underutilized in the global uprising against the coronavirus pandemic? Nanomedicine (Lond). 2020 Jul;15(17):1719-1734. doi: 10.2217/nnm-2020-0163. Epub 2020 May 28. PMID 32462968
- See also: World Health Organization. Coronavirus disease (COVID-19) pandemic. — http://www.who.int/emergencies/diseases/novel-coronavirus-2019